CLINICAL TRIAL: NCT03338361
Title: Efficacy of Approach Avoidance and Attentional Bias Retraining in Alcohol-dependent Patients: a Randomized Controlled Trial in a Clinical Setting
Brief Title: Research on the Efficacy of the "T.O.P. Computer Training" Procedure in the Treatment of Alcohol Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: PZ Heilig Hart (Unknown); PZ Sint-Camillus (Unknown); University of Amsterdam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC/2017/1079
Record Dates: First submitted 2017-10-25; First posted 2017-11-09 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Alcohol Dependence
Keywords: approach avoidance training; attentional bias training; alcohol depencence; relapse
MeSH Terms: conditions — Alcoholism; Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AAT active - VPT sham (Experimental): Approach avoidance training active intervention and visual probe training sham intervention
  Interventions: Behavioral: active approach avoidance training and sham visual probe training
- VPT active - AAT sham (Experimental): Visual probe training active condition and approach avoidance training sham condition
  Interventions: Behavioral: sham approach avoidance training and active visual probe training
- AAT active - VPT active (Experimental): Approach avoidance training active condition and visual probe training active condition
  Interventions: Behavioral: active approach avoidance training and active visual probe training
- AAT sham - VPT sham (Sham Comparator): Approach avoidance training sham condition and visual probe training sham condition
  Interventions: Behavioral: sham approach avoidance training and sham visual probe training

INTERVENTIONS:
Behavioral: active approach avoidance training and sham visual probe training — patients receive active AAT training and sham VPT training
  Arms: AAT active - VPT sham
Behavioral: sham approach avoidance training and active visual probe training — patients receive sham AAT training and active VPT training
  Arms: VPT active - AAT sham
Behavioral: active approach avoidance training and active visual probe training — patients receive active AAT training and active VPT training
  Arms: AAT active - VPT active
Behavioral: sham approach avoidance training and sham visual probe training — patients receive sham AAT training and sham VPT training
  Arms: AAT sham - VPT sham

SUMMARY:
The investigators evaluate the efficacy of a computerised program (T.O.P. tool) consisting of an approach avoidance training (AAT) (to retrain action tendencies for alcohol-related stimuli), a visual probe training (VPT) (to retrain attentional bias for alcohol-related stimuli) and the combination of both training procedures versus placebo training, as an add-on to treatment as usual (psycho-education and cognitive behavioral therapy).

The investigators include hospitalized detoxified alcohol-dependent patients, who receive a four week training procedure, existing of a pre-assessment, 6 training sessions and a post-assessment.

Outcome measures consist of behavioral measures (consumption of alcohol - self report over 1 year), questionnaires (AUDIT; craving on 9-point likert scale) and approach avoidance and visual probe measurement tasks.

A six month and 1 year follow-up is included (behavioral measures and AUDIT). Further, the investigators will also assess credibility (9-point likert scale) of the training procedure before the start of the training and immediately after the assessment of the AAT and VPT training.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized alcohol-dependent patients, choosing for abstinence en committed to treatment
* detoxification (with benzodiazepines) is terminated
* Dutch speaking

Exclusion Criteria:

* neurological condition, such as Korsakoff syndrome
* cognitive problems (cut-off <26/30 on the Montral Cognitive Assessment)
* psychotic disorders
* visual and motor problems at the hands
* non-Dutch speaking
* mental retardation
* patients who are illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
change in drink behavior | baseline, at 6 months and 1-year post training: change in auditscores between baseline, 6 months and 1-year post-training, and differences between groups
  AUDIT score

SECONDARY OUTCOMES:
change in Retraining attentional bias | baseline and between 1 and 7 days after completion of the 6 training sessions: change
  The effect on a VPT task
change in Retraining action tendencies | baseline and between 1 and 7 days after completion of the 6 training sessions: change in action tendencies
  The effect on a AAT task

OTHER OUTCOMES:
change in drinking behavior | baseline; At 3 months post-training: change in audit-c score at baseline and 3 months post training
  score of AUDIT-c (first 3 questions of the AUDIT)
Time to first drink | assessed at 3 months post-training
  Time it takes between finalization of the training and the day the patients drinks an alcoholic beverage
Time to first drink | assessed at 6 months post-training
  Time it takes between finalization of the training and the day the patients drinks an alcoholic beverage
Time to first drink | assessed at 1 year post-training
  Time it takes between finalization of the training and the day the patients drinks an alcoholic beverage
Time to first heavy drinking day | assessed at 3 months post-training
  Time it takes between finalization of the training and the day a female patient drinks ≥ 4 alcoholic units/day and a male patient drinks ≥ 5 alcoholic units/day
Time to first heavy drinking day | assessed at 6 monthspost-training
  Time it takes between finalization of the training and the day a female patient drinks ≥ 4 alcoholic units/day and a male patient drinks ≥ 5 alcoholic units/day
Time to first heavy drinking day | assessed at 1 year post-training
  Time it takes between finalization of the training and the day a female patient drinks ≥ 4 alcoholic units/day and a male patient drinks ≥ 5 alcoholic units/day

CONTACTS AND LOCATIONS:
Overall Officials: sarah C herremans, PhD, MD, Principal Investigator — UZ Gent
Locations (1):
- University Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided